CLINICAL TRIAL: NCT03524105
Title: Promoting Success for Pre-K Teachers, Families and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-01812
Record Dates: First submitted 2018-04-11; First posted 2018-05-14 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Emotional Stress
Keywords: Socio Economic Adversity; Child Development; Poverty; racial disparity; ethnic disparity
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrive Professional Learning plus ParentCorps (Active Comparator)
  Interventions: Behavioral: Program for Parents (Parenting Program)
- Thrive Professional Learning track (Active Comparator)
  Interventions: Behavioral: Thrive Professional Learning

INTERVENTIONS:
Behavioral: Program for Parents (Parenting Program) — Program for Parents (Parenting Program) is implemented by a mental health professional and offered to groups of ~15 parents during the school day and during after school hours. The Program for Parents includes 2-hour sessions provided weekly over a 4-month period. The Program for Students (Friends School Social Emotional Learning Program) is implemented by classroom teachers in the classroom with 90 minute lessons and activities once a week for 14 weeks
  Arms: Thrive Professional Learning plus ParentCorps
Behavioral: Thrive Professional Learning — Professional Learning is delivered to teachers in groups of 20-40 4 times a year over a two-year period. Professional Learning is delivered to leaders in groups of 20 - 40 three times a year over the same two-year period.
  Arms: Thrive Professional Learning track

SUMMARY:
The current study examines the impact of ParentCorps in high-poverty Early Education Centers in New York City (NYC). The study is conducted within the context of the NYC Department of Education (DOE) Pre-K Thrive initiative. As part of this initiative, the Center for Early Childhood Health and Development (CEHD) at NYU Langone Health is implementing services to strengthen family engagement and support parents and teachers in building safe, nurturing and predictable environments for young children. Services include resources to support social emotional learning (SEL) and family engagement (FE) for all Pre-K for All (PKFA) programs and all PKFA families; Professional Learning to support the use of evidence-based SEL and FE practices for teachers and leaders from 350 PKFA programs; and ParentCorps programs for PKFA children and families in 50 PKFA programs (which is a subset of PKFA programs receiving Professional Learning). The current study evaluates the relative value of Thrive Professional Learning plus ParentCorps compared to Thrive Professional Learning.

This study will include 158 pre-K teachers (teachers and teaching assistants) across 23 Centers (12 Centers receiving Thrive Professional Learning plus ParentCorps, 11 Centers receiving Thrive Professional Learning only). All teachers in the 23 Centers will be invited to complete 2 self-report surveys over a two-year period. A sub-set of teachers will be randomly selected to participate in 2 interviews during this period. In addition, teachers in sites randomized to ParentCorps (12 Centers) will be invited to consent to the use of weekly implementation surveys, observational data and semi-structured interviews about experiences with implementation, collected as part of standard implementation practice of ParentCorps, for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Teachers who are teaching staff in the Pre-K classrooms in the 23 Centers.

Exclusion Criteria:

* Only Pre-K teachers from the 23 Centers will be invited to participate in the study. Leaders and other school staff from the Centers are excluded from the study.
* Family-level administrative data only on Pre-K families from the 12 Centers assigned to the Professional Learning plus ParentCorps condition will be obtained from the NYC DOE. Families in other sites are excluded from the request for family-level administrative data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Teacher's knowledge measured using self- report surveys | 15 Months
Teachers' social emotional competencies measured using the Emotion Regulation Questionnaire (ERQ) | 15 Months
  The emotion regulation questionnaire is designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression on a 5 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Brotman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data. To gain access, data requestors will need to sign a data access agreement.